CLINICAL TRIAL: NCT00461617
Title: Multicentre, Double-Dummy, Randomized, Double-Blind Comparison Between Mitiglinide and Nateglinide in the Patients With Type 2 Diabetes
Brief Title: Double-Blind Comparison Between Mitiglinide and Nateglinide in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Gao Xin/Professor, Zhongshan Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAD1301
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes
Keywords: diabetes; rapid and short acting insulin secretagogue; α-glucosidase inhibitor; HbA1C; insulin
MeSH Terms: conditions — Diabetes Mellitus; Fasting; Insulin Resistance | interventions — mitiglinide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator): Nateglinide 120 mg TID
  Interventions: Drug: Mitiglinide

INTERVENTIONS:
Drug: Mitiglinide — 10mg tablet, 10mg TID
  Other Names: Glufast

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Mitiglinide compared to Nateglinide for the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with inadequate control of blood glucose with diet and/or exercise therapy

Exclusion Criteria:

* Type 1 diabetes patients
* Patients who require treatment with insulin
* Patients with severe diabetic complications (neuropathy, retinopathy or nephropathy)
* Patients with severe ketosis, diabetic coma or precoma
* Patients complicated with severe hepatic diseases
* Patients complicated with severe renal diseases
* Patients complicated with severe hypertension
* Patients complicated with severe cardiac disease
* Pregnant women or women possible to be pregnant, nursing women, or women who want to become pregnant during the study period

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1C) | -2, 0, 4, 8, 10, 12, 16, 20 week

SECONDARY OUTCOMES:
Fasting plasma glucose level (FPG) | 0, 4, 8, 12, 16, 20 week
Two-hour postprandial glucose level (PPG2) | 0, 12, 20 week
One-hour postprandial glucose level (PPG1) | 0, 12, 20 week

CONTACTS AND LOCATIONS:
Overall Officials: Xin Gao, Professor, Principal Investigator — Endocrinology Dept. of Fudan University Zhongshan Hospital